CLINICAL TRIAL: NCT00401908
Title: Factors Contributing To Cardiovascular Morbidity and Mortality in Patients With Gastrointestinal Bleeding
Status: Withdrawn | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Ting-Hui Hsieh, Resident Physician, Maimonides Medical Center
Other Study IDs: 06-09-VA02
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Gastrointestinal Bleeding; Acute Coronary Syndrome
Keywords: Acute gastrointestinal bleeding; Acute coronary syndrome
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The rate of complication and death of patients with acute digestive tract bleeding is increased in the setting of acute coronary heart disease. The aim of the study is to establish the relative importance of the risk factors contributing to the death rate from acute digestive tract bleeding in patients admitted with acute coronary heart disease.

DETAILED DESCRIPTION:
The rate of complication and death of patients with acute digestive tract bleeding is increased in the setting of acute coronary heart disease. The aim of the study is to establish the relative importance of the risk factors contributing to the death rate from acute digestive tract bleeding in patients admitted with acute coronary heart disease. This study will be conducted at MMC and involve collecting your clinical information from our medical records and computer systems. Approximately 200 adult patients with acute coronary heart disease and acute digestive tract bleeding admitted to MMC will be enrolled and followed up for 1 year after recruitment. We propose to develop criteria and a scoring system that will assist your doctors in caring for patients like you in the future.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with acute CS and acute GI bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Li, MD, Study Director — Maimonides Medical Center; Scott M Tenner, MD, Principal Investigator — Maimonides Medical Center; Jacob Shani, MD, Principal Investigator — Maimonides Medical Center; Ting-Hui Hsieh, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States